CLINICAL TRIAL: NCT04193826
Title: The Conformal Prague Study: An Evaluation of the Safety and Performance of the Conformal Left Atrial Appendage Seal for Left Atrial Appendage Occlusion
Brief Title: The Conformal Prague Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Conformal Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-101
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Non-valvular Atrial Fibrillation
MeSH Terms: interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Non-valvular AF adults (Experimental): Left atrial appendage closure (LAAC) with the Conformal LAAC device will be performed according to the device Instructions for Use, based on ICE and angiographic guidance, femoral venous access and inter-atrial septum crossing.
  Interventions: Device: Left Atrial Appendage Closure

INTERVENTIONS:
Device: Left Atrial Appendage Closure — Closure of the left atrial appendage (LAAC) is performed percutaneously. Implantation of the LAAC device will be performed according to device specific instructions for use based on both TEE guidance, ICE and angiography, femoral access and inter-atrial septum crossing

SUMMARY:
A prospective, single center, open-label, single arm, study to evaluate the safety and technical performance of the CLAAS system for closure of the left atrial appendage.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate feasibility of ICE as primary imaging modality for device success in patients with non-valvular atrial fibrillation at increased risk for stroke and systemic embolism who are recommended for oral anticoagulation (OAC) therapy but have an appropriate rationale to seek a non-pharmacological alternative to OAC. TEE will be used to confirm the ICE evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female aged ≥18 years
2. Documented non-valvular AF (paroxysmal, persistent, or permanent)
3. High risk of stroke or systemic embolism, defined as a CHA2DS2-VASc score of ≥ 2
4. The patient is recommended for oral anticoagulation therapy (OAC), but has an appropriate rationale to seek a non-pharmacologic alternative to chronic oral anticoagulation
5. The patient is willing and able to comply with the protocol-specified medication regimen and follow-up evaluations
6. The patient (or legally authorized representative) has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent approved by the appropriate Ethics Committee (EC)

Exclusion Criteria:

1. Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following the index procedure. Female patients of childbearing potential must have a negative pregnancy test (per site standard test) within 7 days prior to index procedure.
2. Anatomic conditions that would prevent performance of an LAA occlusion procedure (e.g., prior atrial septal defect [ASD] or patent foramen ovale [PFO], surgical repair or implanted closure device, or obliterated or ligated left atrial appendage)
3. Atrial fibrillation that is defined by a single occurrence or that is transient or reversible (e.g., secondary thyroid disorders, acute alcohol intoxication, trauma, recent major surgical procedures)
4. Patients with a medical condition (other than atrial fibrillation) that mandates chronic oral anticoagulation (e.g., history of unprovoked deep vein thrombosis or pulmonary embolism, or mechanical heart valve)
5. History of bleeding diathesis or coagulopathy, or patients in whom antiplatelet and/or anticoagulant therapy is contraindicated
6. Active infection with bacteremia
7. Documented symptomatic carotid artery disease (>50% diameter stenosis with prior ipsilateral stroke or TIA) or known asymptomatic carotid artery disease (diameter stenosis of >70%)
8. Recent (within 30 days of index procedure) or planned (within 60 days post-procedure) cardiac or non-cardiac interventional or surgical procedure
9. Recent (within 90 days of index procedure) stroke, transient ischemic attack
10. Recent myocardial infarction within 60 days of index procedure
11. Vascular access precluding delivery of implant with catheter-based system
12. Severe heart failure (New York Heart Association Class III or IV)
13. Prior cardiac transplant, history of mitral valve replacement or transcatheter mitral valve intervention, or any mechanical valve implant
14. Renal insufficiency, defined as estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 (by the Modification of Diet in Renal Disease equation), or dialysis at the time of screening
15. Platelet count <100,000 cells/mm3 or >700,000 cells/mm3, or white blood cell count <3,000 cells/mm3
16. Patient has a known allergy, hypersensitivity or contraindication to aspirin, heparin, clopidogrel, prasugrel, ticagrelor, or device materials (e.g., nickel, titanium, gold), or the patient has contrast sensitivity that cannot be adequately pre-medicated
17. Current participation in another investigational drug or device study that interferes with this study
18. Patient is a prisoner
19. Known other medical illness or known history of substance abuse that may cause non-compliance with the protocol or protocol-specified medication regimen, confound the data interpretation, or is associated with a life expectancy of less than 1 year
20. Patient has a condition which precludes adequate transesophageal echocardiographic (TEE) assessment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-19 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Na Homolce, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turagam MK, Neuzil P, Hala P, Mraz T, Dukkipati SR, Reddy VY. Intracardiac Echocardiography-Guided Left Atrial Appendage Closure With a Novel Foam-Based Conformable Device: Safety and 1-Year Outcomes. JACC Clin Electrophysiol. 2022 Feb;8(2):197-207. doi: 10.1016/j.jacep.2021.10.001. Epub 2021 Nov 24. PMID 35210077

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Valvular A-fib Adults: Twenty (20) adult participants with non-valvular atrial fibrillation were assessed and consented to the trial.
Period: Overall Study
Arm/Group | Non-Valvular A-fib Adults
Started | 20
Screen Failed | 1
Implanted | 19
Subject Death | 2
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Participants met the eligibility criteria, consented, and had a procedure attempt.
Arm/Group | Non-valvular AF Adults
Number analyzed (Participants) | 19
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 72.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Czechia | 19

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Major Adverse Events
Description: Major adverse events defined as: All cause mortality, ischemic stroke, systemic thromboembolism, device or procedure-related adverse events requiring open cardiac surgery or major endovascular intervention.
Time Frame: 7 days post-procedure
Measure: Count of Participants; unit: Participants
Groups:
- 7 Day Success: All subjects who had a safety event within 7 days of the successful procedure.
Arm/Group | 7 Day Success
Number analyzed (Participants) | 19
Participants | 19

2. Primary Outcome: Closure Success
Description: Closure success, defined as device success followed by complete closure or peri-device residual leak ≤5 mm in width
Time Frame: 45-days post-procedure
Measure: Count of Participants; unit: Participants
Groups:
- LAA Seal at 45 Days: Breakdown of the seal rate for participants who completed their 45 Day Imaging visit.
Arm/Group | LAA Seal at 45 Days
Number analyzed (Participants) | 15
Participants
  No residual flow | 12
  1 - 2 mm | 3
  >2mm | 0

ADVERSE EVENTS:
Time Frame: 12 Months
Groups:
- Study Adverse Event Breakdown: All site-reported adverse events.
Arm/Group | Study Adverse Event Breakdown
All-Cause Mortality (participants affected / at risk) | 2/19
Serious Adverse Events (participants affected / at risk) | 6/19
Other Adverse Events (participants affected / at risk) | 7/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Adverse Event Breakdown (N=19)
Rapid Ventricular Rate (Cardiac disorders) | 2 (3) — Dyspnea with RVR
Pericardial Effusion (Cardiac disorders) | 2 (2)
Pulmonary Edema (Cardiac disorders) | 1
Device Related Thrombus (Cardiac disorders) | 1
Loss of Consciousness (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Adverse Event Breakdown (N=19)
UTI (Infections and infestations) | 2
Tachyarrhythmia (Cardiac disorders) | 1
Migrating Pain - Head, Chest, Abd (General disorders) | 1
Epistaxis (General disorders) | 1
Headaches (General disorders) | 1
SQ Hematomas (General disorders) | 1
Vomiting (Surgical and medical procedures) | 1
Pericardial Effusion (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT04193826/Prot_SAP_000.pdf